CLINICAL TRIAL: NCT01002872
Title: The Effect of Lanthanum Carbonate on Fibroblast Growth Factor 23 (FGF23 ) in Chronic Kidney Disease
Brief Title: The Effect of Lanthanum Carbonate on Fibroblast Growth Factor 23 ( FGF23) in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Stuart Sprague, Chief, Division of Nephrology and Hypertension Professor of Medicine University of Chicago Medical School, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EH 09-156
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Metabolic Bone Disease
Keywords: FGF23; CKD; Fosrenol; Hyperphosphatemia
MeSH Terms: conditions — Bone Diseases, Metabolic; Hyperphosphatemia | interventions — lanthanum carbonate; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lanthanum Carbonate (Fosrenol) (Active Comparator): Subjects will receive the study drug Lanthanum Carbonate ( Fosrenol)
  Interventions: Drug: Lanthanum Carbonate (Fosrenol)
- Placebo (Placebo Comparator): Subject will receive placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Lanthanum Carbonate (Fosrenol) — Randomization To either Lanthanum Carbonate 1 pill TID/Placebo 1 pill three times a day (TID) Day 15 If phosphorus is 3.5mg/dL-5.5mg/dL Continue with 1 pill TID. If phosphorus <3.5mg/dL Reduce to 1 pill twice a day (BID). If Phosphorus >5.5mg/dL 1 pill with breakfast 1 pill with lunch 2 pills with dinner Day 30 If phosphorus is 3.5mg/dL-5.5mg/dL Continue with 1 pill TID If phosphorus is <3.5mg/dL Reduce to 1 pill daily. If phosphorus >5.5mg/dL 1 pill with breakfast 2 pills with lunch 2 pills with dinner Day 45 If phosphorus is 3.5mg/dL-5.5mg/dL Continue with 1 pill TID If phosphorus <3.5mg/dL stop the drug If phosphorus is >5.5mg/dL 2 pills with breakfast 2 pills with lunch 2 pills with dinner
  Other Names: Fosrenol
  Arms: Lanthanum Carbonate (Fosrenol)
Drug: placebo — Initial dose of placebo will be 1 pill three times a day
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The aim of the study is to assess the effects of the drug lanthanum carbonate (a phosphorus binder drug) on c-terminal and on FGF23 levels in patients with Chronic Kidney Disease (CKD).

Targeting FGF23 measurement in CKD patients may impact both the progression of kidney disease and patient mortality.

DETAILED DESCRIPTION:
This is a double blind randomized placebo controlled pilot study. Subjects with Chronic Kidney Disease ( CKD) stages 3-5 who are not undergoing renal replacement therapy and have not been started on phosphate binders will be randomized to either lanthanum carbonate 1500 mg daily or placebo for a 60 day treatment period. Patient doses will be increased up to a maximum dose of 3000 mg if the serum phosphate is greater than 5.5 mg/dL.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant females ages 18 years of age or older
* Estimated glomerular filtration rate (GFR) between 15-60 ml/min/1.73m
* Serum phosphate > 3.5 mg/dL
* Fibroblast growth factor 2 (FGF2) > 100 relative units per milliliter (RU/mL)
* Corrected serum calcium >8.0mg/dL

Exclusion Criteria:

* Current use of a phosphate binder
* Corrected serum calcium <8.0mg/dL
* Current use of prescription-based vitamin D therapy
* Acute kidney injury in last 3 months
* Significant GI disorder
* History of allergic reaction or sensitivity to lanthanum carbonate
* History of non compliance with visits or medications that preclude study compliance in the opinion of the investigator
* Pregnant or able to become pregnant and unwilling to use a birth control method considered reliable by the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-10; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M Sprague, DO, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be compiled into a manuscript

REFERENCES:
- [Background] Stubbs JR, Quarles LD. Fibroblast growth factor 23: uremic toxin or innocent bystander in chronic kidney disease? Nephrol News Issues. 2009 May;23(6):33-4, 36-7. PMID 19534362
- [Background] Saji F, Shiizaki K, Shimada S, Okada T, Kunimoto K, Sakaguchi T, Hatamura I, Shigematsu T. Regulation of fibroblast growth factor 23 production in bone in uremic rats. Nephron Physiol. 2009;111(4):p59-66. doi: 10.1159/000210389. Epub 2009 Apr 1. PMID 19339809
- [Background] Ibrahim S, Rashed L. Serum fibroblast growth factor-23 levels in chronic haemodialysis patients. Int Urol Nephrol. 2009;41(1):163-9. doi: 10.1007/s11255-008-9466-0. Epub 2008 Oct 7. PMID 18839328
- [Background] Moe SM, Chen NX, Seifert MF, Sinders RM, Duan D, Chen X, Liang Y, Radcliff JS, White KE, Gattone VH 2nd. A rat model of chronic kidney disease-mineral bone disorder. Kidney Int. 2009 Jan;75(2):176-84. doi: 10.1038/ki.2008.456. Epub 2008 Sep 17. PMID 18800026
- [Background] Fliser D, Kollerits B, Neyer U, Ankerst DP, Lhotta K, Lingenhel A, Ritz E, Kronenberg F; MMKD Study Group; Kuen E, Konig P, Kraatz G, Mann JF, Muller GA, Kohler H, Riegler P. Fibroblast growth factor 23 (FGF23) predicts progression of chronic kidney disease: the Mild to Moderate Kidney Disease (MMKD) Study. J Am Soc Nephrol. 2007 Sep;18(9):2600-8. doi: 10.1681/ASN.2006080936. Epub 2007 Jul 26. PMID 17656479
- [Background] Fukagawa M, Kazama JJ. FGF23: its role in renal bone disease. Pediatr Nephrol. 2006 Dec;21(12):1802-6. doi: 10.1007/s00467-006-0230-3. Epub 2006 Aug 24. PMID 16932898

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The date of recruitment 10/27/09-3/7/12.The subjects were seen at Evanston and Glenbrook outpatient clinics
Pre-assignment Details: Subjects who were naive to phosphate binders were enrolled
Period: Overall Study
Arm/Group | Lanthanum Carbonate (Fosrenol) | Placebo
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lanthanum Carbonate (Fosrenol): Subjects will receive the study drug Lanthanum Carbonate ( Fosrenol)
  Lanthanum Carbonate (Fosrenol): Randomization To either Lanthanum Carbonate 1 pill TID/Placebo 1 pill TID Day 15 If phosphorus is 3.5mg/dL-5.5mg/dL Continue with 1 pill TID. If phosphorus <3.5mg/dL Reduce to 1 pill BID. If Phosphorus >5.5mg/dL 1 pill with breakfast 1 pill with lunch 2 pills with dinner Day 30 If phosphorus is 3.5mg/dL-5.5mg/dL Continue with 1 pill TID If phosphorus is <3.5mg/dL Reduce to 1 pill daily. If phosphorus >5.5mg/dL 1 pill with breakfast 2 pills with lunch 2 pills with dinner Day 45 If phosphorus is 3.5mg/dL-5.5mg/dL Continue with 1 pill TID If phosphorus <3.5mg/dL stop the drug If phosphorus is >5.5mg/dL 2 pills with breakfast 2 pills with lunch 2 pills with dinner
- Total: Total of all reporting groups
Arm/Group | Lanthanum Carbonate (Fosrenol) | Placebo | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 5 | 4 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Fibroblast Growth Factor (FGF) 23 Mean Change From Baseline
Description: Mean change from baseline of FGF23 in subjects treated with Lanthanum Carbonate verse placebo at 60 days
Time Frame: Baseline, 60 days
Population: Only patients with readings at both timepoints (baseline and 60 days) were included.
Measure: Mean (Standard Deviation); unit: RU/mL
Arm/Group | Lanthanum Carbonate (Fosrenol) | Placebo
Number analyzed (Participants) | 7 | 6
RU/mL | -62.96 (55.17) | 9.08 (53.84)
Statistical Analysis 1: Comparison: Lanthanum Carbonate (Fosrenol) vs Placebo; Test type: Superiority; p = 0.037, t-test, 2 sided

2. Secondary Outcome: Calcium Mean Change From Baseline
Description: Mean change from baseline Calcium level at 60 days
Time Frame: Baseline, 60 days
Population: Only patients with readings at both timepoints (baseline and 60 days) were included.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lanthanum Carbonate (Fosrenol) | Placebo
Number analyzed (Participants) | 8 | 8
mg/dL | 0.15 (0.49) | 0.04 (0.72)
Statistical Analysis 1: Comparison: Lanthanum Carbonate (Fosrenol) vs Placebo; Test type: Superiority; p = 0.721, t-test, 2 sided

3. Secondary Outcome: Serum Phosphate Mean Change From Baseline
Description: Mean change from baseline serum phosphate at 60 days
Time Frame: Baseline, 60 days
Population: Only patients with readings at both timepoints (baseline and 60 days) were included.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lanthanum Carbonate (Fosrenol) | Placebo
Number analyzed (Participants) | 8 | 8
mg/dL | 0.18 (0.93) | 0.22 (0.54)
Statistical Analysis 1: Comparison: Lanthanum Carbonate (Fosrenol) vs Placebo; Test type: Superiority; p = 0.897, t-test, 2 sided

4. Secondary Outcome: Change From Baseline Serum Parathyroid Hormone
Description: Change from baseline serum parathyroid hormone at 60 days
Time Frame: Baseline, 60 days
Population: Only patients with readings at both timepoints (baseline and 60 days) were included.
Measure: Mean (Standard Deviation); unit: percent change in PTH
Arm/Group | Lanthanum Carbonate (Fosrenol) | Placebo
Number analyzed (Participants) | 8 | 8
percent change in PTH | -18.75 (25.91) | -33.25 (117.70)
Statistical Analysis 1: Comparison: Lanthanum Carbonate (Fosrenol) vs Placebo; Test type: Superiority; p = 0.743, t-test, 2 sided

5. Secondary Outcome: 1,25 Dihydroxyvitamin D 3 Mean Change From Baseline
Description: Mean change from baseline 1,25 dihydroxyvitamin D 3 at 60 days
Time Frame: Baseline, 60 days
Population: Only patients with readings at both timepoints (baseline and 60 days) were included.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lanthanum Carbonate (Fosrenol) | Placebo
Number analyzed (Participants) | 4 | 5
ng/mL | -1.25 (8.66) | -12.20 (23.83)
Statistical Analysis 1: Comparison: Lanthanum Carbonate (Fosrenol) vs Placebo; Test type: Superiority; p = 0.416, t-test, 2 sided

6. Secondary Outcome: 25 Hydroxyvitamin D Mean Change From Baseline
Description: Mean change from baseline 25 hydroxyvitamin D at 60 days
Time Frame: Baseline, 60 days
Population: Only patients with readings at both timepoints (baseline and 60 days) were included.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lanthanum Carbonate (Fosrenol) | Placebo
Number analyzed (Participants) | 7 | 8
ng/mL | 0.43 (6.16) | 2.00 (7.67)
Statistical Analysis 1: Comparison: Lanthanum Carbonate (Fosrenol) vs Placebo; Test type: Superiority; p = 0.672, t-test, 2 sided

7. Secondary Outcome: Serum Alkaline Phosphatase Mean Change From Baseline
Description: Mean change from baseline serum alkaline phosphatase at 60 days
Time Frame: Baseline, 60 days
Population: Only patients with readings at both timepoints (baseline and 60 days) were included.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Lanthanum Carbonate (Fosrenol) | Placebo
Number analyzed (Participants) | 8 | 9
U/L | -0.50 (4.51) | -0.40 (1.91)
Statistical Analysis 1: Comparison: Lanthanum Carbonate (Fosrenol) vs Placebo; Test type: Superiority; p = 0.955, t-test, 2 sided

8. Secondary Outcome: Serum Osteocalcin Mean Change From Baseline
Description: Mean change from baseline serum osteocalcin at 60 days
Time Frame: Baseline, 60 days
Population: Osteocalcin concentrations were not measured
Arm/Group | Lanthanum Carbonate (Fosrenol) | Placebo
Number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Lanthanum Carbonate (Fosrenol) vs Placebo; Test type: Superiority; p < 0.05, t-test, 2 sided

9. Secondary Outcome: 24 Hour Urine Phosphate Mean Change From Baseline
Description: Mean change from baseline 24 hour urine phosphate at 60 days
Time Frame: Baseline, 60 days
Population: Only patients with readings at both timepoints (baseline and 60 days) were included.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Lanthanum Carbonate (Fosrenol) | Placebo
Number analyzed (Participants) | 7 | 6
mg | -148.6 (64.3) | 5.2 (78.7)
Statistical Analysis 1: Comparison: Lanthanum Carbonate (Fosrenol) vs Placebo; Test type: Superiority; p = 0.0066, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | Lanthanum Carbonate (Fosrenol) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 1/10 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanthanum Carbonate (Fosrenol) (N=10) | Placebo (N=9)
mild (General disorders) | 1 (1) | 0 (0) — Broken tooth

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No